CLINICAL TRIAL: NCT06294990
Title: Klinefelter Syndrome - the Effect of Testosterone Treatment in Puberty. a Randomized, Double-blind Placebo-controlled Intervention Study: 'The TiPY Study'
Brief Title: Klinefelter Syndrome and Testosterone Treatment in Puberty
Acronym: TiPY
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Lise Aksglæde (Other)
Responsible Party: Sponsor-Investigator, Lise Aksglæde, Principal investigator, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-505854-16-00
Record Dates: First submitted 2024-02-21; First posted 2024-03-06 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Klinefelter Syndrome
Keywords: Klinefelter syndrome; Puberty; Body composition
MeSH Terms: conditions — Klinefelter Syndrome | interventions — Testosterone

STUDY DESIGN:
Intervention Model Description: Multi-center, national, randomized, double-blind, placebo-controlled intervention study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Testosterone (Active Comparator): Testosterone gel applied to the skin
  Interventions: Drug: Testosterone gel
- Placebo (Placebo Comparator): Placebo gel applied to the skin
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Testosterone gel — Two years treatment with testosterone
  Other Names: Testosterone
  Arms: Testosterone
Other: Placebo — Two years treatment with placebo
  Other Names: Testosterone
  Arms: Placebo

SUMMARY:
The goal of this randomized clinical trial is to study the effect of testosterone replacement therapy during puberty in boys with Klinefelter syndrome (KS, 47,XXY).

The main questions to answer are how treatment with testosterone will affect body fat mass, lipid and glucose metabolism, growth and body proportions, bone mineralization as well as effects on neurocognitive development and emotional and social difficulties.

Participants will be randomized to two years treatment with testosterone or placebo.

DETAILED DESCRIPTION:
Klinefelter syndrome (KS, 47,XXY) is the most frequent sex chromosome disorder with a prevalence of 1:660 boys. Patients with KS are hypogonadal due to a progressive testicular destruction starting already in childhood. Consequently, the adult male with KS is characterized by small testes, signs of incomplete virilization (e.g. lack of voice deepening, sparse face and body hair, gynecomastia, low muscle mass, reduced penile length), hypergonadotropic hypogonadism, infertility and increased risk of metabolic syndrome, diabetes, cardiovascular disease, osteoporosis and psychosocial and neurodevelopmental challenges. Adults with KS have a poor health and a prevention of the major co-morbidities associated with KS and thereby an improvement in the general health would have an enormous impact on the life of a large cohort of males worldwide.

Sufficient testosterone is not only important in the adult but also during puberty and adolescence for a normal virilization and to improve body composition and body proportions, as well as to maximize peak bone mass acquisition. It has therefore been internationally accepted and makes biological sense to consider testosterone replacement therapy (TRT) during puberty in KS. However, there are no evidence based recommendations, and during recent years TRT in puberty has been questioned and is no longer recommended in some countries. There is a need on an international level for evaluating the effect of this treatment. We therefore aim at evaluating the effect of 2 years TRT during early puberty in boys with KS aged 10 to 14 years in this national, multi-center, randomized, double-blind, placebo-controlled intervention study. The primary endpoint is to evaluate the effect on body fat mass. The secondary endpoints are to evaluate effects on lipid and glucose metabolism, growth and body proportions, bone mineralization as well as effects on neurocognitive development and emotional and social difficulties.

ELIGIBILITY:
Inclusion Criteria:

* 47,XXY Klinefelter syndrome
* Age 10-14 years at inclusion
* Luteinizing Hormone > +2 standard deviations (SD) by ultrasensitive luteinizing hormone assay
* Free Testosterone<+2 standard deviations
* Signed consent from parents

Exclusion Criteria:

* Previous or ongoing T treatment except for TRT because of micropenis
* Contraindications to testosterone treatment known hypersensitivity to testosterone or to any other constituent of the gel known or suspected prostatic cancer or breast carcinoma
* Participation in any other clinical trial

Ages: 10 Years to 14 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in body fat mass | Baseline and 1 and two years
  Evaluation of body fat percentage by whole body dual energy x-ray absorptiometry (DEXA) scan

SECONDARY OUTCOMES:
Pubertal development and virilization | Every three months for two years
  Tanner genital (G) staging from G1 to G5. G1 is the prepubertal stage and G5 is the fully develloped stage.
Pubertal development and virilization | Every three months for two years
  Tanner pubic hair (PH) staging from PH1 to PH6. PH1 is the prepubertal stage and PH6 is the fully develloped stage.
Pubertal development and virilization | Every three months for two years
  Measurement of voice frequency using the app "Voice Analyst" (Speechtools Ltd.).
Pubertal development and virilization | Every three months for two years
  Evaluation of testicular volume by palpation with orchidometer
Pubertal development and virilization | Every three months for two years
  Presence of gynecomastia (yes/no)
Pubertal development and viriliztion | Every three months for two years
  Measurement of luteinizing hormone (LH) (IU/L) in serum
Pubertal development and viriliztion | Every three months for two years
  Measurement of serum concentration of testosterone (nmol/L)
Pubertal development and viriliztion | Every three months for two years
  Measurement of folliclestimulating hormone (FSH) (IU/L) in serum
Pubertal development and viriliztion | Every three months for two years
  Measurement of serum concentration of estradiol (pmol/L)
Pubertal development and viriliztion | Every three months for two years
  Measurement of serum concentration of inhibin B (ng/L)
Pubertal development and viriliztion | Every three months for two years
  Measurement of serum concentration of anti mullerian hormone (AMH) (pmol/L)
Pubertal development | At base line, and at 1 and 2 years
  Measurement of the concentration of luteinizing hormone (LH) and follicle stimulating hormone (FSH) in the first, fasting, morning voiding. Measured in IU/L.
Anthropometry | Every three months for two years
  Measurement of height (cm)
Anthropometry | Every three months for two years
  Measurement of weight (kg)
Anthropometry | Every three months for two years
  Measurement of sitting height (cm)
Anthropometry | At base line, and at 1 and 2 years
  Measurement of head circumference (cm)
Anthropometry | At base line, and at 1 and 2 years
  Measurement of arm span (cm)
Bone health | At baseline and at 1 and two years
  Measurement of whole body bone mineral content (BMC) evaluated by whole body DXA scan
Bone health | At base line, and at 1 and 2 years
  Evaluation of bone health index (BHI) from X-ray of left hand and evaluated using the software BoneXpert version 3 (Hørsholm, Denmark)
Measurement of bone turnover markers | At base line, and at 1 and 2 years
  Measurement of 25-OH-vitamin D in blood sample
Measurement of bone turnover markers | At base line, and at 1 and 2 years
  Measurement of calcium in blood sample
Measurement of bone turnover markers | At base line, and at 1 and 2 years
  Measurement of phosphate in blood sample
Measurement of bone turnover markers | At base line, and at 1 and 2 years
  Measurement of parathyroid hormone (PTH) in blood sample
Measurement of bone turnover markers | At base line, and at 1 and 2 years
  Measurement of carboxy terminal telopeptide of collagen type I (CTX) in blood sample
Measurement of bone turnover markers | At base line, and at 1 and 2 years
  Measurement of alkaline phosphatase in blood sample
Measurement of bone turnover markers | At base line, and at 1 and 2 years
  Measurement of osteocalcin in blood sample
Measurement of bone turnover markers | At base line, and at 1 and 2 years
  Measurement of procollagen type I N-terminal peptide (PINP) in blood sample
Changes in growth | Base line and at 1 and 2 years
  Evaluation of bone age by X-ray of left hand and evaluated using the software BoneXpert version 3 (Hørsholm, Denmark)
Measurement of serum concentrations of growth factors | At base line, and at 1 and 2 years
  Measurement of IGF1, IGF2, IGF1BP-1-6 and acid-labile subunit (ALS)) (microg/L)
Muscle strength | Every three months for two years
  Measurement of standing jump length (cm)
Muscle strength | Every three months for two years
  Measurement of hand grip strength using a digital hand dynamometer (Baseline BIMS, digital hand dynamometer, functional model)
Changes i QTc | Base line and at 1 and 2 years
  Evaluation of QT Interval with electrocardiogram (ECG)
Changes in markers of lipids | Base line and at 1 and 2 years
  Measurement of cholesterol in blood sample
Changes in markers of metabolism | Base line and at 1 and 2 years
  Measurement of adiponectin in blood sample
Changes in markers of metabolism | Base line and at 1 and 2 years
  Measurement of leptin in blood sample
Changes in markers of metabolism | Base line and at 1 and 2 years
  Measurement of glucose in blood sample
Changes in markers of metabolism | Base line and at 1 and 2 years
  Measurement of insulin in blood sample
Changes in markers of metabolism | Base line and at 1 and 2 years
  Measurement of HbA1C in blood sample
Changes in markers of inflammation | Base line and at 1 and 2 years
  Measurement of CRP in blood sample
Neuropsychological evaluation | Baseline and after two years
  The Weschler Intelligence Scale for Children - Fifth Edition (WISC-V). The result is based on a combination of seperate index scores. A higher score generally indicates stronger cognitive abilities.
Neuropsychological evaluation | Baseline and after two years
  The Test of Variables of Attention, version 9 (T.O.V.A) is a computerized, performance-based assessment tool used to measure attention and impulsivity. The result is based on a combination of scores.
Neuropsychological evaluation | Baseline and after two years
  The Test of Memory and Learning, Second Edition (Tomal-2). The results are presented as standard scores, scaled scores, percentile ranks, and index scores. A higher score is a better outcome.
Neuropsychological evaluation | Baseline and after two years
  The Judgement of Line Orientation Test. The result is based on a combination of scores. Higher scores indicate better visual-spatial judgment.
Neuropsychological evaluation | Baseline and after two years
  The Mental Rotation Test
Neuropsychological evaluation | Baseline and after two years
  The Beery-Buktenica Developmental Test of Visual-Motor Integration
Neuropsychological evaluation | Baseline and after two years
  The Baseline Speed subtask of the Amsterdam Neuropsychological Tasks program (ANT)
Neuropsychological evaluation | Baseline and after two years
  The Children's Communication Checklist (CCC-2). The result is evaluated based on 10 subscores. Higher scores indicate stronger communication skills.
Neuropsychological evaluation | Baseline and after two years
  The Social Responsiveness Scale-2 (SRS-2) is a standardized questionnaire used to assess social behavior and autism-related traits. Higher scores indicate greater social difficulties, while lower scores suggest stronger social skills.
Neuropsychological evaluation | Baseline and after two years
  The Delis-Kaplan Executive Function System (D-KEFS). Higher scores indicate better executive functioning, while lower scores may suggest difficulties with problem-solving, impulse control, or flexibility.
Neuropsychological evaluation | Baseline and after two years
  The Behavior Rating Inventory of Executive Function, Second Edition rating scale , parent version (BRIEF-2) assesses executive functioning. The result is based on a combination of scores. Higher scores indicate greater executive function difficulties.
Neuropsychological evaluation | Baseline and after two years
  Behavior Assessment System for Children, Third Edition (BASC-3), parent and self-report version. The result is based on a combination of scores. A higher score indicates more difficulties.
Neuropsychological evaluation | Baseline and after two years
  Self-report version of The Multidimensional Anxiety Scale for Children - 2nd edition (MASC-2). The result is based on a combination of scores. Higher scores suggest greater levels of anxiety and more severe symptoms.
Neuropsychological evaluation | Baseline and after two years
  The parent version of the ADHD-rating scale. The result is based on a combination of scores. Higher scores on the inattention and hyperactivity/impulsivity subscales suggest more significant ADHD symptoms.
Neuropsychological evaluation | Baseline and after two years
  The Adaptive Behavior Assessment System, Third Edition (ABAS-III) is a comprehensive tool used to assess adaptive functioning. The result is based on a combination of scores. A higher score indicates better adaptive functioning.
Neuropsychological evaluation | Baseline and after two years
  The Beck Youth Self-Concept Inventory is a tool designed to assess self-concept and self-esteem in children and adolescents. A high percentile rank (above 70) indicates a strong self-concept, while a low percentile rank (below 30) suggests low self-esteem or dissatisfaction.
Neuropsychological evaluation | Baseline and after two years
  PedsQL Multidimentional Fatigue Scale, parent, and self-report versions is a tool designed to assess fatigue levels in children and adolescents. The result is based on a combination of scores. A higher score indicates less fatigue (better energy levels and functioning). A lower score indicates more fatigue, suggesting that fatigue is significantly affecting the child's daily activities.
Cryopreservation of spermatozoa | After 2 years
  If the patient is able and willing he will have the possibility to deliver a semen sample for cryopreservation of potential spermatozoa
Epigenetic | At base line, and at 1 and 2 years
  The effects on epigenetics will be evaluation by evaluating changes in DNA methylation patterns. This will be analyzed on DNA from white blood cells by applying Illumina methylation arrays.
Genetic effects | At base line, and at 1 and 2 years
  DNA will be analyzed using a selected set of genetic polymorphisms in target genes with established or theoretic effects on hormone production and hormone receptor sensitivity. They will be analysed either by PCR genotyping or targeted sequencing (max. 200 selected genes). SNP arrays that exclusively target common variants, and not any rare variants, will be used to determine the influence of common genetic variation on the observed associations.
Small non-coding RNA | At base line, and at 1 and 2 years
  RNA analysis of circulating, small, non-coding RNA will be performed as a biomarker for the circulating concentrations of reproductive hormones and for overweight.

CONTACTS AND LOCATIONS:
Overall Officials: Lise Aksglaede, MD, Principal Investigator — Copenhagen University Hospital, Rigshospitalet, Copenhagen, Denmark
Locations (1):
- Copenhagen University Hospital, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Caspersen ID, Fritzboger AFO, Petersen JH, Birkebaek N, Christensen AR, Schou AJ, Kristensen K, Ross JL, Davis S, Butler G, van Rijn S, Juul A, Aksglaede L. Effect of testosterone treatment during puberty in boys with Klinefelter syndrome (The TIPY Study): protocol for a nationwide randomised, double-blinded, placebo-controlled study. BMJ Open. 2025 Mar 15;15(3):e095628. doi: 10.1136/bmjopen-2024-095628. PMID 40090688